CLINICAL TRIAL: NCT01615614
Title: A Phase I, Open-Label Study in Healthy Subjects, to Explore the Pharmacokinetics of Different Dosing Regimens of Rilpivirine in Combination With Rifabutin, at Steady-State
Brief Title: A Study to Explore the Pharmacokinetics of Rilpivirine With Rifabutin in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen R&D Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR100812; TMC278IFD1003 (Other: Janssen R&D Ireland); 2012-000141-12 (EudraCT Number)
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-03

CONDITIONS: Healthy
Keywords: Rilpivirine; Rifabutin; Pharmacokinetics; Healthy participants
MeSH Terms: interventions — Rilpivirine; Rifabutin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental): Rilpivirine 25 mg once daily will be administered for 11 days
  Interventions: Drug: Rilpivirine
- Treatment B (Experimental): Rilpivirine 50 mg once daily will be administered for 11 days and rifabutin 300 mg once daily will be administered for 17 days
  Interventions: Drug: Rilpivirine; Drug: Rifabutin
- Treatment C (Experimental): Rilpivirine (in a regimen to be determined based on an interim pharmacokinetic analysis of treatment A and B) will be administered for 11 days and rifabutin 300 mg once daily will be administered for 17 days.
  Interventions: Drug: Rilpivirine; Drug: Rifabutin

INTERVENTIONS:
Drug: Rilpivirine — Type=exact number, unit=mg, number=25, 50, and will be determined after treatment A and B analysis form=tablet, route=oral. Once or twice daily with a total daily dose of rilpivirine between 25 and 75 mg will be administered for 11 days.
Drug: Rifabutin — Type=exact number, unit=mg, number=150, form=capsule, route=oral. Two capsules daily will be administered for 17 days.
  Arms: Treatment B; Treatment C

SUMMARY:
The purpose of this study is to explore the pharmacokinetics of different dosing regimens of rilpivirine in combination with rifabutin in healthy participants.

DETAILED DESCRIPTION:
This is a Phase I, open-label (the participant will know the identity of the treatment they receive), 3-period study to investigate the pharmacokinetic (what the body does to the medication) interaction of steady-state (constant concentrations in your blood resulting from a fixed dosing regimen) rilpivirine and steady-state rifabutin. Twenty healthy participants will be enrolled and will receive 3 different treatments (treatment A: rilpivirine 25 mg once daily administered daily for 11 days; treatment B: rilpivirine 50 mg once daily administered for 11 days + rifabutin 300 mg daily administered for 17 days; treatment C: rilpivirine (in a regimen to be determined based on an interim analysis of treatments A and B) administered for 11 days + rifabutin 300 mg daily administered for 17 days). All 20 participants will be randomized (the study drug is assigned by chance) to receive treatments A (10 participants) and treatment B (10 participants) and there will be a washout period of at least 21 days between treatments A and B. After all participants have completed treatments A and B, there will be an interim analysis to decide upon the dosing regimen for rilpivirine in treatment C (the rilpivirine regimen in treatment C could be either once daily or twice daily with a total daily dose of rilpivirine between 25 and 75 mg). All 20 participants will receive treatment C. Safety and tolerability will be evaluated throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants should be healthy on the basis of physical examination, medical history, vital signs, electrocardiogram, and the results of blood biochemistry and hematology tests and a urinalysis performed at screening
* Men must agree to use a highly effective method of birth control (ie, male condom with either female intrauterine device, diaphragm, cervical cap or hormone based contraceptives by their female partner), and to not donate sperm during the study and for 3 months after receiving the last dose of study drug
* Women must be postmenopausal for at least 2 years, or be surgically sterile (have had a total hysterectomy or bilateral oophorectomy, tubal ligation/bilateral tubal clips without reversal operation, or otherwise be incapable of becoming pregnant)
* Women must have a negative pregnancy test at screening
* Participants must be non-smoking for at least 3 months prior to screening

Exclusion Criteria:

* A positive HIV-1 or HIV-2 test at screening
* History or suspicion of alcohol or barbiturate, amphetamine, recreational or narcotic drug use which in the Investigator's opinion would compromise subject safety and/or compliance with study procedures
* Hepatitis A, B or C infection (confirmed by hepatitis A IgM, HBsAg, or hepatitis C virus antibody, respectively) at screening
* Currently active clinically significant gastrointestinal, cardiovascular, neurologic, psychiatric, metabolic, endocrine, renal, hepatic, respiratory, inflammatory or infectious disease
* Any history of tuberculosis, ocular herpes, or uveitis
* Currently significant diarrhea or gastric stasis that in the Investigator's opinion could influence drug absorption or bioavailability

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of different dosing regimens of rilpivirine in combination with rifabutin, at steady-state | Up to 168 hours (postdose)
  Pharmacokinetics of different dosing regimens of rilpivirine in combination with rifabutin, at steady-state will be evaluated.

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | Up to 87 days
  Number of participants with adverse events will be evaluated to assess safety and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Merksem, Belgium